CLINICAL TRIAL: NCT05346107
Title: PLD Plus Cyclophosphamide Followed by Nab-paclitaxel (Nab-P) as Primary Chemotherapy Continuously Combined With Dual HER2 Blockage for HER2-positive Breast Cancer: A Single-arm Phase 2 Trial(Brecan Trial)
Brief Title: PLD-cyclophosphamide-Nab-P Continuously Combined With Dual HER2 Blockage for HER2-positive Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20223267-1
Record Dates: First submitted 2022-03-28; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; 1-dodecylpyridoxal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PldCHP---Nab-PHP (Experimental): he patients were treated with PldCHP (pegylated liposomal doxorubicin 35mg/m2, cyclophosphamide 600mg/m2, trastuzumab 8 mg/kg loading, then 6 mg/kg, pertuzumab 840 mg loading, then 420 mg, iv, q3w) for 4 cycles followed by Nab-PHP (Nab-Paclitaxel 260mg/m2, trastuzumab 6 mg/kg, pertuzumab 420 mg, iv, q3w) for 4 cycles, with strict monitoring of cardiotoxicity.
  Interventions: Drug: pegylated liposomal doxorubicin (PLD) plus cyclophosphamide followed by Nab-paclitaxel (Nab-P) ,continuously combined with dual HER2 blockage

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin (PLD) plus cyclophosphamide followed by Nab-paclitaxel (Nab-P) ,continuously combined with dual HER2 blockage — The patients were treated with PldCHP (pegylated liposomal doxorubicin 35mg/m2, cyclophosphamide 600mg/m2, trastuzumab 8 mg/kg loading, then 6 mg/kg, pertuzumab 840 mg loading, then 420 mg, iv, q3w) for 4 cycles followed by Nab-PHP (Nab-Paclitaxel 260mg/m2, trastuzumab 6 mg/kg, pertuzumab 420 mg, iv, q3w) for 4 cycles, with strict monitoring of cardiotoxicity.

SUMMARY:
patients with HER2-positive breast cancer (cT2-3/N0-1/M0) were treated with PldCHP (pegylated liposomal doxorubicin 35mg/m2, cyclophosphamide 600mg/m2, trastuzumab 8 mg/kg loading, then 6 mg/kg, pertuzumab 840 mg loading, then 420 mg, iv, q3w) for 4 cycles followed by Nab-PHP (Nab-Paclitaxel 260mg/m2, trastuzumab 6 mg/kg, pertuzumab 420 mg, iv, q3w) for 4 cycles

DETAILED DESCRIPTION:
Upon approval by the Medical Ethics Committee of Xijing Hospital, patients with HER2-positive breast cancer (cT2-3/N0-1/M0) receiving neoadjuvant therapy, were enrolled. The patients were treated with PldCHP (pegylated liposomal doxorubicin 35mg/m2, cyclophosphamide 600mg/m2, trastuzumab 8 mg/kg loading, then 6 mg/kg, pertuzumab 840 mg loading, then 420 mg, iv, q3w) for 4 cycles followed by Nab-PHP (Nab-Paclitaxel 260mg/m2, trastuzumab 6 mg/kg, pertuzumab 420 mg, iv, q3w) for 4 cycles, with strict monitoring of cardiotoxicity. The primary endpoint was pCR rate, and secondary endpoints were cardiac safety during neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. HER2-positive breast cancer
2. cT2-3/N0-1/M0
3. aged18-80 years
4. receiving neoadjuvant therapy
5. ECOGPS score 0 or 1
6. Able to understand the test requirements, willing and able to comply with the test and follow-up procedures
7. Adequate organ function

Exclusion Criteria:

1. cardiac, hepatic, renal, or psychiatric disease history
2. History of other malignancy within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of pathological complete response | At the end of Cycle 1 (each cycle is 14 days)
  absence of invasive carcinoma in the breast and axillary lymph nodes, while residual ductal carcinoma in situ was accepted (ypT0orTisypN0)

SECONDARY OUTCOMES:
adverse effects | during the period of neadjuvant chemotherapy, an average of 14 days
  Serious adverse effect occur within neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital ， Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang JX, Yang YQ, Hu WY, Yang L, Wu J, Wen XX, Yu J, Huang ML, Xu DD, Tie DC, Wang L, Li FF, Li NL. A Phase II Study of Neoadjuvant PLD/Cyclophosphamide and Sequential nab-Paclitaxel Plus Dual HER2 Blockade in HER2-Positive Breast Cancer. Oncologist. 2024 Jan 5;29(1):e15-e24. doi: 10.1093/oncolo/oyad160. PMID 37279780